CLINICAL TRIAL: NCT05622955
Title: A Novel Approach to Endometriosis Treatment: Piloting an Interdisciplinary Group Care Model
Brief Title: Endometriosis Group Care
Acronym: PEEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202206202
Record Dates: First submitted 2022-11-10; First posted 2022-11-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Group care; Integrative care; Pelvic floor physical therapy; Yoga; Mindfulness; Patient-centered outcomes
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometriosis group care (Experimental): Groups of 6-10 patients with endometriosis and chronic pelvic pain will attend eight weekly two-hour sessions.
  Interventions: Other: Peer Empowered Endometriosis Pain Support (PEEPS)

INTERVENTIONS:
Other: Peer Empowered Endometriosis Pain Support (PEEPS) — The sessions will provide education on endometriosis, mindfulness, yoga, nutrition, and strategies to cope with chronic pain. Patients will additionally receive peer and clinician support to decrease the social isolation experienced by people with endometriosis

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the Peer Empowered Endometriosis Pain Support (PEEPS) program in people living with endometriosis-related pelvic pain. The main question[s] it aims to answer are:

* Is PEEPS effective at decreasing pain interference and improving patient-reported quality of life outcomes?
* What are the barriers and facilitators to PEEPS implementation? Participants will engage in eight weekly 2-hour sessions led by an endometriosis specialist, pain psychologist, pelvic floor physical therapist, and yoga instructor. At these sessions they will participate in peer support, education, mindfulness, and yoga.

DETAILED DESCRIPTION:
This is an 8 week interdisciplinary, integrative group care program conducted through the Department of Obstetrics and Gynecology (OB/GYN) at Washington University in St. Louis (WUSTL). The program, called PEEPS, incorporates mindfulness, physical therapy, yoga, physical activity, nutrition, and education. Additionally, PEEPS will provide peer support and demonstrate investment of individual clinicians and the healthcare system.

The program focuses on equipping participants with pain management and coping skills so they have an expanded toolkit to manage their pain after completing the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-48 years
* Operative confirmation of endometriosis
* Chronic pelvic pain (defined as pain perceived to originate from the pelvis, lasting ≥6 months)
* No plan to have surgery in next 12 weeks
* Be able to attend eight 2-hour weekly sessions on the Washington University campus

Exclusion Criteria:

* Non-English speaking
* Currently pregnant
* Severe physical impairment
* History of hip or spine surgery
* Opioid use ≥ 5 days in the past 3 months, other than for the 6-week post-operative period
* Current or history of psychiatric disorder with psychosis
* Vulvadynia or vaginismus

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pain Interference | 8 weeks
  Change in reported pain after PEEPS program completion by Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference

SECONDARY OUTCOMES:
Physical Function | 8 weeks
  Change in reported physical function, measured by the PROMIS Physical Function Scale
Sexual Function | 8 weeks
  Change in reported sexual function, measured by the Female Sexual Function Index
Endometriosis-specific quality of life | 8 weeks
  Endometriosis-specific quality of life, measured by Endometriosis Health Profile-30
Anxiety | 8 weeks
  Change in reported anxiety, measured by the PROMIS Anxiety Scale
Depression | 8 weeks
  Change in reported depression, measured by the PROMIS Depression Scale
Pain Catastrophizing | 8 weeks
  Change in reported catastrophizing, measured by the Pain Catastrophizing Scale
Overall symptom improvement | 8 weeks
  Change in overall symptoms, measured by the Patient Global Impression of Change Scale
Modified every day discrimination scale | Baseline
  To assess experiences of healthcare discrimination

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mowers EL, Lim CS, Skinner B, Mahnert N, Kamdar N, Morgan DM, As-Sanie S. Prevalence of Endometriosis During Abdominal or Laparoscopic Hysterectomy for Chronic Pelvic Pain. Obstet Gynecol. 2016 Jun;127(6):1045-1053. doi: 10.1097/AOG.0000000000001422. PMID 27159755
- [Background] Missmer SA, Cramer DW. The epidemiology of endometriosis. Obstet Gynecol Clin North Am. 2003 Mar;30(1):1-19, vii. doi: 10.1016/s0889-8545(02)00050-5. PMID 12699255
- [Background] As-Sanie S, Black R, Giudice LC, Gray Valbrun T, Gupta J, Jones B, Laufer MR, Milspaw AT, Missmer SA, Norman A, Taylor RN, Wallace K, Williams Z, Yong PJ, Nebel RA. Assessing research gaps and unmet needs in endometriosis. Am J Obstet Gynecol. 2019 Aug;221(2):86-94. doi: 10.1016/j.ajog.2019.02.033. Epub 2019 Feb 18. PMID 30790565
- [Background] Walker EA, Katon WJ, Hansom J, Harrop-Griffiths J, Holm L, Jones ML, Hickok LR, Russo J. Psychiatric diagnoses and sexual victimization in women with chronic pelvic pain. Psychosomatics. 1995 Nov-Dec;36(6):531-40. doi: 10.1016/S0033-3182(95)71608-5. PMID 7501783
- [Background] Meltzer-Brody S, Leserman J, Zolnoun D, Steege J, Green E, Teich A. Trauma and posttraumatic stress disorder in women with chronic pelvic pain. Obstet Gynecol. 2007 Apr;109(4):902-8. doi: 10.1097/01.AOG.0000258296.35538.88. PMID 17400852
- [Background] Latthe P, Mignini L, Gray R, Hills R, Khan K. Factors predisposing women to chronic pelvic pain: systematic review. BMJ. 2006 Apr 1;332(7544):749-55. doi: 10.1136/bmj.38748.697465.55. Epub 2006 Feb 16. PMID 16484239
- [Background] Fourquet J, Sinaii N, Stratton P, Khayel F, Alvarez-Garriga C, Bayona M, Ballweg ML, Flores I. Characteristics of women with endometriosis from the USA and Puerto Rico. J Endometr Pelvic Pain Disord. 2015 Oct-Dec;7(4):129-135. doi: 10.5301/je.5000224. Epub 2015 Oct 1. PMID 27331050
- [Background] Delanerolle G, Ramakrishnan R, Hapangama D, Zeng Y, Shetty A, Elneil S, Chong S, Hirsch M, Oyewole M, Phiri P, Elliot K, Kothari T, Rogers B, Sandle N, Haque N, Pluchino N, Silem M, O'Hara R, Hull ML, Majumder K, Shi JQ, Raymont V. A systematic review and meta-analysis of the Endometriosis and Mental-Health Sequelae; The ELEMI Project. Womens Health (Lond). 2021 Jan-Dec;17:17455065211019717. doi: 10.1177/17455065211019717. PMID 34053382
- [Background] Falcone T, Flyckt R. Clinical Management of Endometriosis. Obstet Gynecol. 2018 Mar;131(3):557-571. doi: 10.1097/AOG.0000000000002469. PMID 29420391
- [Background] Williams AC, Eccleston C, Morley S. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007407. doi: 10.1002/14651858.CD007407.pub3. PMID 23152245
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Smith CA, Armour M, Zhu X, Li X, Lu ZY, Song J. Acupuncture for dysmenorrhoea. Cochrane Database Syst Rev. 2016 Apr 18;4(4):CD007854. doi: 10.1002/14651858.CD007854.pub3. PMID 27087494
- [Background] Monticone M, Ambrosini E, Rocca B, Cazzaniga D, Liquori V, Pedrocchi A, Vernon H. Group-based multimodal exercises integrated with cognitive-behavioural therapy improve disability, pain and quality of life of subjects with chronic neck pain: a randomized controlled trial with one-year follow-up. Clin Rehabil. 2017 Jun;31(6):742-752. doi: 10.1177/0269215516651979. Epub 2016 May 31. PMID 27246516 (Retraction: PMID 36069340 Clin Rehabil. 2022 Nov;36(11):1423)
- [Background] van Koulil S, van Lankveld W, Kraaimaat FW, van Helmond T, Vedder A, van Hoorn H, Donders R, de Jong AJ, Haverman JF, Korff KJ, van Riel PL, Cats HA, Evers AW. Tailored cognitive-behavioral therapy and exercise training for high-risk patients with fibromyalgia. Arthritis Care Res (Hoboken). 2010 Oct;62(10):1377-85. doi: 10.1002/acr.20268. PMID 20521308
- [Background] Meissner K, Schweizer-Arau A, Limmer A, Preibisch C, Popovici RM, Lange I, de Oriol B, Beissner F. Psychotherapy With Somatosensory Stimulation for Endometriosis-Associated Pain: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1134-1142. doi: 10.1097/AOG.0000000000001691. PMID 27741200
- [Background] Lemstra M, Olszynski WP. The effectiveness of multidisciplinary rehabilitation in the treatment of fibromyalgia: a randomized controlled trial. Clin J Pain. 2005 Mar-Apr;21(2):166-74. doi: 10.1097/00002508-200503000-00008. PMID 15722810
- [Background] Weijenborg PT, Ter Kuile MM, Gopie JP, Spinhoven P. Predictors of outcome in a cohort of women with chronic pelvic pain - a follow-up study. Eur J Pain. 2009 Aug;13(7):769-75. doi: 10.1016/j.ejpain.2008.09.002. Epub 2008 Oct 16. PMID 18929498
- [Background] Weijenborg PT, Ter Kuile MM, Stones W. A cognitive behavioural based assessment of women with chronic pelvic pain. J Psychosom Obstet Gynaecol. 2009 Dec;30(4):262-8. doi: 10.3109/01674820903378742. PMID 19922399
- [Background] Allaire C, Williams C, Bodmer-Roy S, Zhu S, Arion K, Ambacher K, Wu J, Yosef A, Wong F, Noga H, Britnell S, Yager H, Bedaiwy MA, Albert AY, Lisonkova S, Yong PJ. Chronic pelvic pain in an interdisciplinary setting: 1-year prospective cohort. Am J Obstet Gynecol. 2018 Jan;218(1):114.e1-114.e12. doi: 10.1016/j.ajog.2017.10.002. Epub 2017 Oct 12. PMID 29031895
- [Background] Beaton-Starr M, Rist PM, Connor JP, Wayne PM, Osypiuk K, Bernstein C. Development and Implementation of the Integrative Toolbox for Headache Management. Headache. 2020 Apr;60(4):771-775. doi: 10.1111/head.13743. Epub 2020 Jan 9. PMID 31919834
- [Background] Harpole LH, Samsa GP, Jurgelski AE, Shipley JL, Bernstein A, Matchar DB. Headache management program improves outcome for chronic headache. Headache. 2003 Jul-Aug;43(7):715-24. doi: 10.1046/j.1526-4610.2003.03128.x. PMID 12890125
- [Background] Murphy SE, Blake C, Power CK, Fullen BM. Comparison of a Stratified Group Intervention (STarT Back) With Usual Group Care in Patients With Low Back Pain: A Nonrandomized Controlled Trial. Spine (Phila Pa 1976). 2016 Apr;41(8):645-52. doi: 10.1097/BRS.0000000000001305. PMID 26630423
- [Background] Chao MT, Abercrombie PD, Santana T, Duncan LG. Applying the RE-AIM Framework to Evaluate Integrative Medicine Group Visits Among Diverse Women with Chronic Pelvic Pain. Pain Manag Nurs. 2015 Dec;16(6):920-9. doi: 10.1016/j.pmn.2015.07.007. Epub 2015 Sep 10. PMID 26365760
- [Background] Chao MT, Abercrombie PD, Duncan LG. Centering as a model for group visits among women with chronic pelvic pain. J Obstet Gynecol Neonatal Nurs. 2012 Sep-Oct;41(5):703-10. doi: 10.1111/j.1552-6909.2012.01406.x. Epub 2012 Aug 3. PMID 22862426
- [Background] Mellado BH, Falcone AC, Poli-Neto OB, Rosa E Silva JC, Nogueira AA, Candido-Dos-Reis FJ. Social isolation in women with endometriosis and chronic pelvic pain. Int J Gynaecol Obstet. 2016 May;133(2):199-201. doi: 10.1016/j.ijgo.2015.08.024. Epub 2016 Jan 6. PMID 26873129
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Consolidated Framework for Implmentation Research. https://cfirguide.org/constructs/. Published 2021. Accessed 14 December, 2021
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Damschroder LJ, Reardon CM, Opra Widerquist MA, Lowery J. Conceptualizing outcomes for use with the Consolidated Framework for Implementation Research (CFIR): the CFIR Outcomes Addendum. Implement Sci. 2022 Jan 22;17(1):7. doi: 10.1186/s13012-021-01181-5. PMID 35065675
- [Background] Simoens S, Dunselman G, Dirksen C, Hummelshoj L, Bokor A, Brandes I, Brodszky V, Canis M, Colombo GL, DeLeire T, Falcone T, Graham B, Halis G, Horne A, Kanj O, Kjer JJ, Kristensen J, Lebovic D, Mueller M, Vigano P, Wullschleger M, D'Hooghe T. The burden of endometriosis: costs and quality of life of women with endometriosis and treated in referral centres. Hum Reprod. 2012 May;27(5):1292-9. doi: 10.1093/humrep/des073. Epub 2012 Mar 14. PMID 22422778
- [Background] Soliman AM, Yang H, Du EX, Kelley C, Winkel C. The direct and indirect costs associated with endometriosis: a systematic literature review. Hum Reprod. 2016 Apr;31(4):712-22. doi: 10.1093/humrep/dev335. Epub 2016 Feb 6. PMID 26851604
- [Background] Soliman AM, Coyne KS, Gries KS, Castelli-Haley J, Snabes MC, Surrey ES. The Effect of Endometriosis Symptoms on Absenteeism and Presenteeism in the Workplace and at Home. J Manag Care Spec Pharm. 2017 Jul;23(7):745-754. doi: 10.18553/jmcp.2017.23.7.745. PMID 28650252
- [Background] Gupta J, Cardoso LF, Harris CS, Dance AD, Seckin T, Baker N, Ferguson YO. How do adolescent girls and boys perceive symptoms suggestive of endometriosis among their peers? Findings from focus group discussions in New York City. BMJ Open. 2018 Jun 4;8(6):e020657. doi: 10.1136/bmjopen-2017-020657. PMID 29866728
- [Background] Joosten YA, Israel TL, Williams NA, Boone LR, Schlundt DG, Mouton CP, Dittus RS, Bernard GR, Wilkins CH. Community Engagement Studios: A Structured Approach to Obtaining Meaningful Input From Stakeholders to Inform Research. Acad Med. 2015 Dec;90(12):1646-50. doi: 10.1097/ACM.0000000000000794. PMID 26107879
- [Background] Fox SD, Flynn E, Allen RH. Mindfulness meditation for women with chronic pelvic pain: a pilot study. J Reprod Med. 2011 Mar-Apr;56(3-4):158-62. PMID 21542535
- [Background] Rod K. Observing the Effects of Mindfulness-Based Meditation on Anxiety and Depression in Chronic Pain Patients. Psychiatr Danub. 2015 Sep;27 Suppl 1:S209-11. PMID 26417764
- [Background] Andersen TE, Vaegter HB. A 13-Weeks Mindfulness Based Pain Management Program Improves Psychological Distress in Patients with Chronic Pain Compared with Waiting List Controls. Clin Pract Epidemiol Ment Health. 2016 Jun 30;12:49-58. doi: 10.2174/1745017901612010049. eCollection 2016. PMID 27708686
- [Background] Nygaard AS, Rydningen MB, Stedenfeldt M, Wojniusz S, Larsen M, Lindsetmo RO, Haugstad GK, Oian P. Group-based multimodal physical therapy in women with chronic pelvic pain: A randomized controlled trial. Acta Obstet Gynecol Scand. 2020 Oct;99(10):1320-1329. doi: 10.1111/aogs.13896. Epub 2020 Jun 1. PMID 32386466
- [Background] Grinberg K, Weissman-Fogel I, Lowenstein L, Abramov L, Granot M. How Does Myofascial Physical Therapy Attenuate Pain in Chronic Pelvic Pain Syndrome? Pain Res Manag. 2019 Dec 12;2019:6091257. doi: 10.1155/2019/6091257. eCollection 2019. PMID 31915499
- [Background] Huang AJ, Rowen TS, Abercrombie P, Subak LL, Schembri M, Plaut T, Chao MT. Development and Feasibility of a Group-Based Therapeutic Yoga Program for Women with Chronic Pelvic Pain. Pain Med. 2017 Oct 1;18(10):1864-1872. doi: 10.1093/pm/pnw306. PMID 28419385
- [Background] Goncalves AV, Barros NF, Bahamondes L. The Practice of Hatha Yoga for the Treatment of Pain Associated with Endometriosis. J Altern Complement Med. 2017 Jan;23(1):45-52. doi: 10.1089/acm.2015.0343. Epub 2016 Nov 21. PMID 27869485
- [Background] Goncalves AV, Makuch MY, Setubal MS, Barros NF, Bahamondes L. A Qualitative Study on the Practice of Yoga for Women with Pain-Associated Endometriosis. J Altern Complement Med. 2016 Dec;22(12):977-982. doi: 10.1089/acm.2016.0021. Epub 2016 Aug 23. PMID 27552065
- [Background] HealthMeasures. PROMIS Short Form v2.0 - Pain Intensity - 3a. Northwestern University. https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=3379&Itemid= 992. Published 2020. Accessed 02/09/2022
- [Background] Innovation OU. Endometriosis Health Profile-30 (EHP-30). https://innovation.ox.ac.uk/outcome- measures/endometriosis-health-profile-ehp/. Published 2016. Accessed 02/09/2022.
- [Background] HealthMeasures. PROMIS Short Form v2.0 - Physical Function 10a. Northwestern University. https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=794&Itemid=9 92. Published 2020. Accessed 02/09/2022.
- [Background] HealthMeasures. PROMIS Short Form v1.0 - Anxiety - 7a. Northwestern University. https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=146&Itemid=9 92. Published 2016. Accessed 02/09/2022.
- [Background] HealthMeasures. PROMIS Short Form v1.0 Depression - 8b. Northwestern University. https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=157&Itemid=9 92. Published 2016. Accessed 02/09/2022.
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Sullivan MJ. The Pain Catastrophizing Scale User Manual. McGill University. https://aspecthealth.ca/wp-content/uploads/2017/03/PCSManual_English1.pdf. Published 2009. Accessed 02/09/2022.
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Williams DR, Yan Yu, Jackson JS, Anderson NB. Racial Differences in Physical and Mental Health: Socio-economic Status, Stress and Discrimination. J Health Psychol. 1997 Jul;2(3):335-51. doi: 10.1177/135910539700200305. PMID 22013026
- [Background] Whitehead AL, Sully BG, Campbell MJ. Pilot and feasibility studies: is there a difference from each other and from a randomised controlled trial? Contemp Clin Trials. 2014 May;38(1):130-3. doi: 10.1016/j.cct.2014.04.001. Epub 2014 Apr 13. PMID 24735841
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] CFIR Guide. https://cfirguide.org/guide/app/#/. Published 2022. Accessed 2/6/2022.
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Repository IO. ImplementationOutcomeRepository.org. https://implementationoutcomerepository.org/. Accessed 2/6/2022.
- [Background] Mohamed EA, Giama NH, Shaleh HM, Kerandi L, Oseini AM, Ahmed Mohammed H, Kerandi H, Allotey LK, Waaeys IA, Ali HA, Ali HM, Mohamed SA, Yang JD, Gaga WO, Tamire LL, Windissa A, Patten CA, Balls-Berry JE, Roberts LR. Knowledge, Attitudes, and Behaviors of Viral Hepatitis Among Recent African Immigrants in the United States: A Community Based Participatory Research Qualitative Study. Front Public Health. 2020 Mar 6;8:25. doi: 10.3389/fpubh.2020.00025. eCollection 2020. PMID 32211358